CLINICAL TRIAL: NCT02450305
Title: Hyperbaric Oxygen and Its Effect on Radiation Induced Long Term Side Effects
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Marvin Heyboer, MD, State University of New York - Upstate Medical University
Other Study IDs: 482428 HBO
Record Dates: First submitted 2015-05-18; First posted 2015-05-21 (Estimated); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Cancer of Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treated with HBO: QOL questionnaires at 5 time points for those having HBO therapy at least one year post radiation therapy for head and neck cancer, daily x6 weeks
- Not treated with HBO: QOL questionnaires for those at least one year post radiation therapy for head and neck cancer at 5 times points.

SUMMARY:
The investigators intend to determine if patients that are already undergoing Hyperbaric Oxygen (HBO) therapy one year post treatment with radiation therapy for head and neck cancer, experience improvement in xerostomia and/or taste alteration. The investigators will enroll a similar demographic one year post treatment with radiation therapy that does not receive HBO therapy. This is a quality of life study.

DETAILED DESCRIPTION:
Radiation therapy is a commonly utilized treatment modality for head and neck cancer patients. Xerostomia (i.e. dry mouth) (and taste change) are common and most significant side effects of this treatment. Xerostomia leads to several complications for patients including difficulty in chewing, speaking, swallowing, taste and smell abnormalities, oral infections and inflammation, osteoradionecrosis, dental caries and periodontal disease. These conditions tend to lead to an overall decreased quality of life for patients affected.

A possible modality for the treatment of xerostomia is the use of hyperbaric oxygen (HBO) therapy. HBO is the medical use of oxygen at a level higher than atmospheric pressure. It has been proposed that HBO results in accelerated blood vessel growth and repair in tissue injuries by increasing the oxygen partial pressure gradient (Bennett, 2005). Today, the use of HBO is widely accepted for both the treatment and prevention of radiation induced toxicities such as osteoradionecrosis and soft tissue necrosis.

Here at Upstate University Hospital, the investigators treat approximately 20 patients each year with hyperbaric oxygen for either the prevention or management of radiation induced complications such as osteoradionecrosis and /or soft tissue necrosis. The investigators would like to use this group of patients to evaluate the effect of HBO in the improvement of radiation induced xerostomia (and or taste change). The investigators' data will be collected from patients with the use of periodic quality of life questionnaires at 5 timepoints, as well as data relating to the treatment each patient was given. .

ELIGIBILITY:
Inclusion Criteria:

* males and females age > 18 previous radiation therapy to the head and neck region at least one year from end of treatment

Exclusion Criteria:

* history of parotidectomy history of dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that will be receiving HBO therapy for head and neck cancer related side effects and matched controls not receiving HBO therapy
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2013-08; Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Xerostomia | one year
  The improvement of xerostomia following HBO therapy will be measured using standard RTOG head and neck cancer questionnaires.

SECONDARY OUTCOMES:
Taste alteration | one year
  The improvement of taste alteration following HBO therapy will be measured using standard RTOG head and neck cancer questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Marvin Heyboer, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No